CLINICAL TRIAL: NCT01049425
Title: Randomised Comparison of Adjuvant Docetaxel / Cyclophosphamide With Sequential Adjuvant EC / Docetaxel Chemotherapy in Patients With HER2/Neu Negative Early Breast Cancer
Brief Title: Anthracycline-free Taxane Based Chemotherapy in Patients With HER2/Neu Negative Early Breast Cancer
Acronym: planB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Sanofi (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG AM04
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Primary Breast Cancer; Her2 Non-overexpressing
Keywords: anthracycline-free; OncotypDX; taxane; Her2 negative breast cancer
MeSH Terms: interventions — Epirubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epirubicin and Cyclophosphamid followed by Docetaxel (Active Comparator): 4 cycles of EC on day one every three weeks followed by 4 cycles of Docetaxel on day one every three weeks
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- Combination of Docetaxel and Cyclophosphamid (Experimental): intravenous infusion on day one every three weeks
  Interventions: Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Epirubicin — 4 cycles, intravenous use, day 1 every three weeks
  Arms: Epirubicin and Cyclophosphamid followed by Docetaxel
Drug: Cyclophosphamide — 4 cycles, intravenous infusion, day 1 every three weeks
  Arms: Epirubicin and Cyclophosphamid followed by Docetaxel
Drug: Docetaxel — 4 cycles, intravenous infusion, day 1 every three weeks after completion of EC-chemotherapy
  Arms: Epirubicin and Cyclophosphamid followed by Docetaxel
Drug: Cyclophosphamide — 6 cycles, intravenous infusion, day 1 every 3 weeks
  Arms: Combination of Docetaxel and Cyclophosphamid
Drug: Docetaxel — 6 cycles, intravenous infusion, day one every three weeks
  Arms: Combination of Docetaxel and Cyclophosphamid

SUMMARY:
The planned trial compares an anthracycline-free taxane based regimen versus a modern third generation (anthracycline/taxane-based) regimen in HER2/neu non-over expressing tumors. The aim is to define a further anthracycline-free standard and to spare anthracycline toxicity to a patient, who will only have a modest benefit from this compound. Prior to randomization for chemotherapy for all patients with HR positive disease OncotypeDX® will be performed to identify patients who should not receive chemotherapy.

Secondary objectives of this trial will be to compare overall survival and toxicity between the two chemotherapy arms, to evaluate survival in the observation arm and to perform translational research regarding prognostic and predictive factors.

ELIGIBILITY:
Inclusion Criteria(Screening):

* Female patients, age at diagnosis 18 - 75 years
* Histological confirmed unilateral primary invasive carcinoma of the breast
* Adequate surgical treatment with complete resection of the tumor (R0) and resection of > or = 10 axillary nodes or SLN in clinically N0 patients
* T1 - T4 (if operable, inflammatory breast cancer is excluded)
* Her-2 non-over expressing tumor confirmed by IHC/FISH
* Estrogen and/or progesterone receptor analysis performed on the primary tumor prior to randomization. Results must be known at the time of randomization
* Node positive disease or node negative disease with at least one other risk factor (tumor size > or = 2 cm, grade > or = 2, ER and PR negative, high uPA//PAI-1 levels)
* No evidence for distant metastasis (M0) after conventional staging
* Performance Status ECOG < or = 1 or KI > or = 80 %
* The patient must be accessible for treatment and follow-up
* Written informed consent for central pathology review and evaluation of Recurrence Score (HR positive) and participation in the planB trial prior to beginning specific protocol procedures

HR positive patients:

* Patient willingness to participate in adjuvant chemotherapy planB trial if RS > 11
* Indication for chemotherapy given provided either > 4 involved lymph nodes or RS > 11 in 1-3 lymph nodes or N0 disease

Additional Inclusion Criteria (Randomisation to chemotherapy):

* Laboratory requirements (within 21 days prior to randomization):

  * Leucocytes > or = 3.5 109/L
  * platelets > or = 100 109/L
  * haemoglobin > or = 10 g/dL
  * total bilirubin < or = 1 ULN
  * ASAT (SGOT) and ALAT (SGPT) < or = 2.5 UNL
  * creatinine < 175 ymol/L (2 mg/dL)
* Negative pregnancy test (urine or serum) within 7 days prior to randomization in premenopausal patients
* LVEF within normal limits of each institution measured by echocardiography or MUGA scan and

Exclusion Criteria(Screening):

* HER2 over expression confirmed by IHC/FISH/CISH
* Known hypersensitivity reaction to the compounds or incorporated substances
* Known polyneuropathy > or = grade 2
* Severe and relevant comorbidity that would interact with the application of cytotoxic agents or the participation in the study including acute cystitis and ischuria and chronic kidney disease.
* Prior malignancy with a disease-free survival of < 10 years, except curatively treated basalioma of the skin, pTis of the cervix uteri or ipsilateral ductal carcinoma in-situ (DCISpTis of the breast)
* Non-operable breast cancer including inflammatory breast cancer
* Previous or concurrent treatment with cytotoxic agents for any reason after consultation with the sponsor
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry
* Male breast cancer
* Concurrent pregnancy; patients of childbearing potential must implement a highly effective (less then 1% failure rate) non-hormonal contraceptive measures during the study treatment
* Breast feeding woman
* Sequential breast cancer
* Lack of patient compliance

Additional Exclusion Criteria (Randomisation):

* Inadequate organ function including:

  * Leucocytes < 3,5 G/l
  * platelets < 100 G/l
  * creatinine or bilirubin above normal limits
  * alkaline phosphatise > 5 UNL
  * ASAT and/or ALAT associated with AP > 2.5 UNL
  * uncompensated cardiac function
* Time since axillary dissection > 42 days

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3198 (Actual)
Dates: Start 2009-02-05 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
disease-free survival in patients treated with either 6 cycles of Docetaxel / Cyclophosphamide chemotherapy or 4 cycles of EC followed by 4 cycles of Docetaxel as adjuvant treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike A. Nitz, Prof. Dr. med., Principal Investigator — Ev. Krankenhaus Bethesda Moenchengladbach; Nadia Harbeck, Prof. Dr. med., Study Chair — University Hospital Cologne
Locations (1):
- Bethesda Krankenhaus, Mönchengladbach, Germany

REFERENCES:
- [Derived] Sechi A, Mijnes J, Villwock S, Rose M, Steib F, Bringezu S, Berger J, Schalla C, von Serenyi S, Dietrich J, Ortiz-Bruchle N, Heij L, Bednarsch J, Gluz O, Nitz U, Harbeck N, Graeser M, Zu Eulenburg C, Mohammadian MP, Jozwiak K, Kreipe HH, Christgen M, Radner M, Jonigk D, Dahl E. The Janus Face of SPAG6: Inducing EMT in Luminal Breast Cancer Cells Amidst Widespread Expression Loss in Breast Tumours. J Cell Mol Med. 2025 Oct;29(19):e70870. doi: 10.1111/jcmm.70870. PMID 41066509
- [Derived] Kolberg-Liedtke C, Gluz O, Heinisch F, Feuerhake F, Kreipe H, Clemens M, Nuding B, Malter W, Reimer T, Wuerstlein R, Graeser M, Shak S, Nitz U, Kates R, Christgen M, Harbeck N. Association of TILs with clinical parameters, Recurrence Score(R) results, and prognosis in patients with early HER2-negative breast cancer (BC)-a translational analysis of the prospective WSG PlanB trial. Breast Cancer Res. 2020 May 14;22(1):47. doi: 10.1186/s13058-020-01283-w. PMID 32408905
- [Derived] Nitz U, Gluz O, Clemens M, Malter W, Reimer T, Nuding B, Aktas B, Stefek A, Pollmanns A, Lorenz-Salehi F, Uleer C, Krabisch P, Kuemmel S, Liedtke C, Shak S, Wuerstlein R, Christgen M, Kates RE, Kreipe HH, Harbeck N; West German Study Group PlanB Investigators. West German Study PlanB Trial: Adjuvant Four Cycles of Epirubicin and Cyclophosphamide Plus Docetaxel Versus Six Cycles of Docetaxel and Cyclophosphamide in HER2-Negative Early Breast Cancer. J Clin Oncol. 2019 Apr 1;37(10):799-808. doi: 10.1200/JCO.18.00028. Epub 2019 Feb 20. PMID 30785826
- [Derived] Nitz U, Gluz O, Christgen M, Kates RE, Clemens M, Malter W, Nuding B, Aktas B, Kuemmel S, Reimer T, Stefek A, Lorenz-Salehi F, Krabisch P, Just M, Augustin D, Liedtke C, Chao C, Shak S, Wuerstlein R, Kreipe HH, Harbeck N. Reducing chemotherapy use in clinically high-risk, genomically low-risk pN0 and pN1 early breast cancer patients: five-year data from the prospective, randomised phase 3 West German Study Group (WSG) PlanB trial. Breast Cancer Res Treat. 2017 Oct;165(3):573-583. doi: 10.1007/s10549-017-4358-6. Epub 2017 Jun 29. PMID 28664507
- [Derived] Gluz O, Nitz UA, Christgen M, Kates RE, Shak S, Clemens M, Kraemer S, Aktas B, Kuemmel S, Reimer T, Kusche M, Heyl V, Lorenz-Salehi F, Just M, Hofmann D, Degenhardt T, Liedtke C, Svedman C, Wuerstlein R, Kreipe HH, Harbeck N. West German Study Group Phase III PlanB Trial: First Prospective Outcome Data for the 21-Gene Recurrence Score Assay and Concordance of Prognostic Markers by Central and Local Pathology Assessment. J Clin Oncol. 2016 Jul 10;34(20):2341-9. doi: 10.1200/JCO.2015.63.5383. Epub 2016 Feb 29. PMID 26926676